CLINICAL TRIAL: NCT03898089
Title: The Effects of Myofascial Release Technique Combined With Core Stabilization Training in Elderly With Non-Specific Low Back Pain
Brief Title: The Effects of Myofascial Release Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Ismail OZSOY, Principal Investigator, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019100
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Low Back Pain; Exercise; Elderly
Keywords: Myofascial Release Technique; Core Stabilization Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Investigator
Masking Description: Single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Exercise Group (Other): The participants in the core stability exercise group will be included in a treatment program for 3 days per week for 6 weeks.
  Interventions: Other: Core Stability Exercise
- Core Exercise plus Myofascial Relaxation Group (Experimental): In addition to the core stabilization exercises myofascial relaxation technique will be performed with roller massager (Theraband®, The Hygenic Corporation, Akron, OH.) for 3 days per week for 6 weeks.
  Interventions: Other: Core Stability Exercise plus Myofascial Release Technique Group

INTERVENTIONS:
Other: Core Stability Exercise — The participants in the core stability exercise group will be included in a treatment program for 3 days per week for 6 weeks. Traditional physiotherapy methods will be applied to all participants. Traditional physiotherapy will include heat modality (a hot pack for 15 minutes), electrotherapy (transcutaneous electrical nerve stimulation (TENS), a 50 Hz conventional TENS with a pulse duration <150 microseconds).Each training session will be lasted 60 min, starting with a 10-min warm up program mainly consisting of core strength exercises and ending with a 5-min cool-down program (stretching). Progression of exercises will be tailored to individual patients' ability, fatigue and pain. Exercises will be designed from 1 set to 3 sets, from 8 to 15 repetitions and contractions from 5 seconds to 10 seconds.
  Arms: Core Exercise Group
Other: Core Stability Exercise plus Myofascial Release Technique Group — In addition to the core stabilization exercise group myofascial relaxation technique will be performed with roller massager (Theraband®, The Hygenic Corporation, Akron, OH.) for 3 days per week for 6 weeks. The myofascial relaxation technique will be performed along the superficial back line (plantar fascia gastrocnemius muscles, hamstring muscles, sacrolumbar fascia, erector spinae muscles) bilaterally. Myofascial relaxation will be done to the anatomical structures indicated by roller massage technique. Applications will be made in 3 sets of 30sec for each zone (1 min rest between sets) and 7/10 according to VAS.
  Arms: Core Exercise plus Myofascial Relaxation Group

SUMMARY:
This study is designed as a single blind randomized controlled trial. Thirty-six elderly with non-specific low back pain (NSLBP) will be recruited. The participants will randomly divided two parallel groups as control and intervention. Traditional physiotherapy methods will be applied to all participants. Traditional physiotherapy will include heat modality (a hot pack for 15 minutes), electrotherapy (transcutaneous electrical nerve stimulation (TENS), a 50 Hz conventional TENS with a pulse duration <150 microseconds). For the control group, core stability exercise will be applied 3 days/week, 6 weeks. For the intervention group, in addition to the core stabilization exercises myofascial relaxation technique will be performed with roller massager ((Thera-Band; The Hygenic Corporation, Akron, OH) 3 days/week, 6 weeks. The myofascial relaxation technique will be performed along the superficial back line. To the best of our knowledge, there is no randomized controlled study investigating the effect of the myofascial release technique combined with core stabilization in elderly with NSLBP. This study aimed to investigate the myofascial release technique combined with core stabilization exercise in elderly with NSLBP.

DETAILED DESCRIPTION:
Low back pain is a symptom that is an important health problem throughout the world. Non-specific low back pain (NSLBP) is the most widespread form of the low back pain. The NSLBP is called low back pain without recognisable specific underlying pathology. The lifetime prevalence of low back pain is up to 84%. The prevalence and burden the low back pain of increases with aging.

The use of various methods of non-pharmacological and non-invasive especially exercise, mobilization, and manipulation in low back pain. Core stability exercise is a common exercise modality in the treatment of low back pain. Core stability exercises improve trunk strength and low back disability in elderly with NSLBP. However, the studies have showed that decreasing strength in the deep muscles (such as the transverse abdominis and multifidus) is accompanied by increased activation in the superficial muscles (such as the erector spina) in patients with low back pain. Therefore, myofascial release technique on superficial muscles can be effective in NSLBP.

To the best of our knowledge, there is no randomized controlled study investigating the effect of the myofascial release technique combined with core stabilization in elderly with NSLBP. Therefore, this study aimed to investigate the myofascial release technique combined with core stabilization exercise in elderly with NSLBP.

ELIGIBILITY:
Inclusion Criteria:

* Ongoing low back pain for at least 3 months
* Having no neurological, rheumatological or musculoskeletal problems
* Standardized Mini-Mental State score greater than or equal to 24 points

Exclusion Criteria:

* Low back pain originating from various pathologies
* Presence of cord compression,
* Radiculopathy,
* Osteoporosis or osteopenia (t score>-1),
* Long-term use of anticoagulant or corticosteroid drugs,
* Patients who had received any treatment for their low back pain.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 weeks
  The visual analog scale is a validated, subjective measure for pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Pain Pressure Threshold | 6 weeks
  An electronic pressure algometer (Algometer commander, JTech Medical, Line; Salt Lake City) is used to measure pressure pain threshold (PPT) with a stimulation surface area of 1 cm2. Three consecutive measurements are performed at each site, with 10 seconds of recovery time allowed between repeated applications. During the algometric measurements, the subjects are asked to say "yes" when the pain is experienced. The amount of pressure-causing pain is recorded as PPT in kg/ cm2. The subjects are required to lie down in a prone position for the measurements. 2 lumbar paravertebral points (bilateral 5 cm lateral to the L3 spinous processes) are evaluated.
The Oswestry Disability Index | 6 weeks
  It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. If a patient marks more than one statement in a question, the highest scoring statement is recorded as a true indication of disability.
Chair Sit and Reach Test | 6 weeks
  Subjects are asked to sit at the edge of a chair with one leg extend forward with knee straight, heel on the floor and ankle bended as 90o , while the other foot remained flat on the floor. Subjects are instructed to place one hand over the other hand with the middle finger tips even, and tried to reach forward to the toe of the extended leg. The distance between the middle finger tips and the toe are recorded.

SECONDARY OUTCOMES:
Supine Bridge Test | 6 weeks
  Subjects are asked to lie down and bend their knees in full contact with the floor of the feet. In this position (hooked position) they are asked to lift their hips from the bed. The time for the bridge is measured in seconds after stopping the contact of the hips with the bed.
Tampa Scale of Kinesiophobia | 6 weeks
  This scale is used to assess the patients' fear of pain or re-injury due to movement. It consists of 17 items and assesses various factors of fear/avoidance and injury/re-injury in several activities. Total score of the scale varies between 17 and 68 and higher scores represent higher levels of kinesiophobia.
Berg Balance Scale | 6 weeks
  The scale consists of 14 items that are scored on a scale of 0 to 4. A score of 0 is given if the participant is unable to do the task, and a score of 4 is given if the participant is able to complete the task based on the criterion that has been assigned to it. The maximum total score on the test is 56. The items include simple mobility tasks (eg transfers, standing unsupported, sit-to-stand) and more difficult tasks.
Spinal Mobility Assessment | 6 weeks
  Assessment of spinal mobility with the Spinal Mouse System (Idiag, Fehraltorf, Switzerland), a hand-held, computer-assisted electromechanical device.
The World Health Organization Quality of Life Instrument-Older Adults Module (WHOQOL-OLD) | 6 weeks
  The WHOQOL-OLD is a questionnaire consisting of 24 items related to 6 different domains: sensorial operation, autonomy, death and dying past, present and future activities, social participation, and intimacy. Each domain includes 4 items, with each individual score ranging from 1 to 5 and the range of possible marks varying from 5 to 20 for all domains. The scores of the 24 WHOQOL-OLD module items are combined to produce a general score, known as the "total score", indicating the senior citizens' quality of life reports, ranging from 24 to 120.
Gait Cycle Assessment | 6 weeks
  Assessment of gait cycle with device (Biodex Gait Trainer 2, Biodex Medical Systems Inc, US). Gait cycle (sec) is determined by walking subjects on the gait trainer for 6 minute.
Walking Speed Assessment | 6 weeks
  Assessment of walking speed with device (Biodex Gait Trainer 2, Biodex Medical Systems Inc, US). Walking speed (m/sec) is determined by walking subjects on the gait trainer for 6 minute.
Maximum Walking Distance Assessment | 6 weeks
  Assessment of maximum walking distance with device (Biodex Gait Trainer 2, Biodex Medical Systems Inc, US). Maximum walking distance (m) is determined by walking subjects on the gait trainer for 6 minute.
Step Length Assessment | 6 weeks
  Assessment of step length with device (Biodex Gait Trainer 2, Biodex Medical Systems Inc, US). Step length (cm) is determined by walking subjects on the gait trainer for 6 minute.
Ambulation Index Assessment | 6 weeks
  Assessment of ambulation index with device (Biodex Gait Trainer 2, Biodex Medical Systems Inc, US). Ambulation index score is determined by walking subjects on the gait trainer for 6 minute.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Ozsoy, PhD, Principal Investigator — Kırşehir Ahi Evran University School of Physical Therapy and Rehabilitation
Locations (1):
- Kırşehir Ahi Evran University School of Physical Therapy and Rehabilitation, Kırşehir, Turkey (Türkiye)

REFERENCES:
- [Derived] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992